CLINICAL TRIAL: NCT00457067
Title: Pilot Study of Intravitreal Injection of Ranibizumab for Macular Telangiectasia With Neovascularization
Brief Title: Injected Ranibizumab to Treat Macular Telangiectasia With New Blood Vessel Formation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070095; 07-EI-0095
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-24

CONDITIONS: Telangiectasia
Keywords: Hyperfluorescence on Fluorescein; Idiopathic Juxtafoveal Telangiectasia; Retinal Edema/Thinning; Vascular Endothelial Growth Factor; Macular Telangiectasia
MeSH Terms: conditions — Telangiectasis; Idiopathic Juxtafoveal Retinal Telangiectasia; Papilledema | interventions — Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab

SUMMARY:
This study will examine whether the drug ranibizumab is an effective treatment for macular telangiectasia, a condition in which existing blood vessels near the macula (the back part of the eye responsible for sharp central vision) become dilated and twisted, and new abnormal blood vessels may form under the retina. Both the existing dilated vessels, as well the new subretinal vessels can leak fluid and blood, distort the retina, and affect vision. This study will see if ranibizumab can slow or stop the leakage and growth of new vessels forming under the retina.

Patients 18 years of age and older who have macular telangiectasia in both eyes and new blood vessel formation under the retina in at least one eye may be eligible for this study. Visual acuity must be 20/40 or worse.

Participants receive at least four injections of ranibizumab into the eye over a 12-week period. After the fourth injection, additional injections may be given every 4 weeks for up to 1 year if the doctor determines that they may be of benefit. In addition to ranibizumab treatment, patients undergo the following procedures:

* Medical history and physical examination.
* Eye examination, including dilation of the pupils and measurement of the fluid pressure in the eye.
* Fluorescein angiogram: A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Photographs of the retina are taken with a special camera that flashes a blue light into the eye. The photos show whether any dye has leaked from the vessels into the retina.
* Indocyanine green angiography: This procedure identifies feeder vessels that may be supplying the abnormal blood vessels. The test is similar to fluorescein angiography, but uses a green dye and flashes an invisible light.
* Autofluorescence imaging: This test examines how well the retina functions. The back of the eye is photographed with a bright light.
* Optical coherence tomography: This test measures retinal thickness. A light shined into the eye produces cross-sectional pictures of the retina. The measurements are repeated during the study to determine if retinal thickening is getting better or worse, or staying the same.
* Stereoscopic color fundus photography: The pupils are dilated and special photographs of the inside of the eye are taken to evaluate the retina and measure changes that occur over time. The camera flashes a bright light into the eye for each picture.
* Follow-up visits: The doctor evaluates the effects of the study treatment before and after each injection. Patients are contacted by phone 3 days after each injection to check on any treatment side effects. A final follow-up visit is scheduled 8 weeks after the last treatment.

DETAILED DESCRIPTION:
Retinal telangiectasis is a group of rare, idiopathic retinal vascular anomalies affecting the retinal capillaries in which irregular capillary dilation and incompetence occur in the macula. This is the former group 2 in the Gass classification of idiopathic juxtafoveal telangiectasia in which fluorescein angiography showed leakage with capillary dilation. These patients typically are diagnosed in their fifth or sixth decade of life. Both sexes may be affected. Minimal exudation, superficial retinal crystalline deposits, and right-angle venules characterize this disorder. As the disease progresses, intraretinal pigment plaques and eventually subretinal/choroidal neovascularization develop. Currently, these patients will be classified as macular telangiectasia. The pathogenesis of the disease is unknown. Because of the leakage of the retinal vessels and also the finding of neovascularization, it is possible that vascular endothelial growth factor (VEGF) may be implicated in this disease.

The purpose of this study is to evaluate the possible role of ranibizumab for the treatment of five participants with macular telangiectasia with hyperfluorescence on fluorescein angiography, with vision decreased to 20/40 or worse, with neovascularization. The primary outcome will be a visual acuity change, either increase or decrease of 15 letters or more at one year. The secondary outcomes measured at one year will include visual acuity changes of 10 letters or more, the change in retinal thickening documented by OCT, the extent and degree of fluorescein leakage, the change in area of hypofluorescence, and the change in central retinal sensitivity. This is a pilot study designed to evaluate the feasibility and potential efficacy of treating patients with macular telangiectasia in a larger, phase III study within the organization of the MAC TEL Research Group, sponsored by the Lowy Foundation. Currently, the research group is enrolling 200 patients affected with this condition for a natural history study in 22 international clinical centers.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participant must understand and sign the informed consent.
  2. Participant must be at least 18 years of age.
  3. Participant must have macular telangiectasia in both eyes.
  4. Participant must have neovascularization in the study eye.
  5. Participant must have vision loss of 20/40 or worse.
  6. Participant must have clear ocular media and adequate papillary dilation to permit good quality stereoscopic fundus photography.
  7. All women of childbearing potential must have a negative urine pregnancy test at baseline, and be willing to undergo testing immediately prior to each injection and monthly for at least 2 months following the last dose of ranibizumab.
  8. Women of child-bearing potential who are sexually active and men who are sexually active are required to use two forms of birth control during the course of the study.

EXCLUSION CRITERIA:

1. History (within past 5 years) or evidence of severe cardiac disease (apparent in electrocardiogram abnormalities, clinical history of unstable angina, acute coronary syndrome, myocardial infarction, revascularization procedure within 6 months prior to baseline, atrial or ventricular tachyarrythmias requiring ongoing treatment).
2. History of stroke within 12 months of study entry.
3. History within the past five years of a chronic ocular or periocular infection (including any history of ocular herpes zoster).
4. Current acute ocular or periocular infection.
5. Any major surgical procedure within one month of study entry.
6. Known serious allergies to fluorescein dye.
7. Previous participation in a clinical trial (for either eye) involving anti-angiogenic drugs (pegaptanib, ranibizumab, bevacizumab, anecortave acetate, Protein Kinase C inhibitors, etc.).
8. Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye.
9. History of vitrectomy surgery in the study eye.
10. History of glaucoma filtering surgery in the study eye.
11. History of corneal transplant in the study eye.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2007-03-27; Study Completion 2007-10-24

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gass JD. Histopathologic study of presumed parafoveal telangiectasis. Retina. 2000;20(2):226-7. doi: 10.1097/00006982-200002000-00028. No abstract available. PMID 10783967